CLINICAL TRIAL: NCT06248775
Title: Nursing Prehabilitation Intervention Supported With Technology for Vascular Surgery in People With Type 2 Diabetes
Acronym: VITAAAL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nicole Oosterom (Other)
Responsible Party: Sponsor-Investigator, Nicole Oosterom, MSc, Ziekenhuisgroep Twente
Organization: Ziekenhuisgroep Twente (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: W2310 0450
Record Dates: First submitted 2023-11-14; First posted 2024-02-08 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Type 2 Diabetes; Lifestyle; Prehabilitation; Vascular Surgery
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Technology; Amyloid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nursing prehabilitation intervention group (Other): Patients all undergo the intervention aimed at lifestyle improvement and glucose regulation
  Interventions: Behavioral: Prehabilitation Intervention Supported with Technology (Fitbit, glucose sensor and app for diet habits)

INTERVENTIONS:
Behavioral: Prehabilitation Intervention Supported with Technology (Fitbit, glucose sensor and app for diet habits) — During the VITAAAL intervention patients use the Diameter app to monitor their physical activities (in connection with a Fitbit), nutrition (using the Diameter app) and glucose levels (in connection with Freestyle Libre 2 sensors). Before the intervention starts, a three-day period of blinded baseline measurements is performed to measure current habits, motivation and possibilities. Then, individual aims for improving vitality are formulated in consultation with the NP diabetes. Afterwards, patients continue measuring their habits unblinded with the Diameter for the following weeks and weekly evaluate their goals with the nurse practitioner to receive new instructions and/or to adapt the goals

SUMMARY:
Type 2 Diabetes Mellitus (T2DM) is the most common chronic lifestyle-related disorder with a significant impact on quality and healthcare expenditures. Insufficient glycemic control and low fitness level prior to a surgical intervention results in more postoperative complications which leads to a longer hospitalization, higher costs and mortality. A prehabilitation intervention in persons with T2DM prior to surgery should be aimed to improve glucose regulation and translate into better outcomes. However, the classic interventions such as Combined Lifestyle Intervention are labor-intensive and require a high degree of organization and therefore are not used as standard care. The use of biofeedback can provide a solution to this. Biofeedback with a continuous glucose sensor in combination with lifestyle monitoring by activity trackers and coaching prior to surgery is a promising but unexplored prehabilitation strategy. The Nursing Prehabilitation Intervention Supported with Technology for vascular Surgery in People with Type 2 Diabetes (VITAAAL) intervention is a form of blended care. It focuses on improving vitality and glycemic control before surgery with the Diameter application, using intermittently scanned glucose monitoring, nutrition habits and physical activity blended with coaching from a nurse practitioner (NP) diabetes. Because VITAAAL is a novel intervention, the aim of this pilot study is to investigate its usability and feasibility. The pilot study consists of three phases. After the first phase, a specific prehabilitation module will be designed and programmed in the Diameter app. This module will be based on the results and experiences in phase one. In phase two and three the patients will use the adjusted version of the Diameter app that contains implemented findings of the previous phase.

ELIGIBILITY:
Inclusion Criteria:

* Patients with T2DM who need a scheduled vascular surgery, consisting of AAA surgery endovascular or classical abdominal approach, aortic stenosis surgery or Fontaine II.
* Aged 18 years or older
* Being familiar with using an Android smartphone (version 5.0 or higher);
* Participant can understand and weigh up information provided by researcher and can understand what the consequences of participation are.

Exclusion Criteria:

* Need for acute vascular surgery
* Dependency on renal replacement therapy
* Known with (pre)proliferative diabetic retinopathy with or without macula oedema.
* Any general diseases or mental disorder rendering participation in the study impossible
* Drug abuse
* Insufficient mastery of the Dutch language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-11-16 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
usability of the VITAAAL intervention | 4 to 8 weeks prior surgery
  Usability will be assessed by means of an open-ended interview. The purpose of the interview is to gain insight into the experiences with the VITAAAL intervention regarding usability to identify user problems. To investigate the usability of the VITAAAL intervention, an interview scheme has been drawn up. The following topics will be discussed: overall experience, learnability, efficiency, memorability, satisfaction, errors and positive and negative elements
Acceptability of the VITAAAL intervention | 4 to 8 weeks prior surgery
  Acceptability will be assessed using the UTAUT2 questionnaire. The UTAUT2 questionnaire consists of 19 questions. The UTAUT2 determinants include performance expectancy, effort expectancy, pleasure/hedonic motivation, facilitating circumstances, design, technical issues and habit. In addition, we will ask about the (potential) contribution of the VITAAAL intervention, the 3 most positive and negative aspects of the VITAAAL intervention and an overall rating expressed in a score on a scale of 1 to 10 (1 = extremely poor, 10 = excellent). The experiences with the VITAAAL intervention will be assessed using multiple statements generated by the research team according to literature and previous used UTAUT2-model based questionnaires. Each statement will be scored on a 7-point Likert scale (1 = extremely disagree, 7 = extremely agree) where a higher score indicate positive experiences with the VITAAAL intervention.

SECONDARY OUTCOMES:
Glycemic regulation - Time in Range | 4 to 8 weeks prior surgery
  Time in Range represents the total time per day that the sensor-measured interstitial glucose concentration is between 3.9 and 10.0 mmol/L assessed with the Freestyle Libre.
Glycemic regulation - Time Above Range (TAR) | 4 to 8 weeks prior surgery
  TAR represents the total time per day that the sensor-measured interstitial glucose concentration value is above 10.0 mmol/L. The TAR will be calculated with algorithms based on the glucose values assessed with the Freestyle Libre.
Glycemic regulation - Time Below Range (TBR) | 4 to 8 weeks prior surgery
  TBR represents the total time per day that the sensor-measured interstitial glucose concentration is below 3.9 mmol/L assessed with the Freestyle Libre.
Glucose management indicator (GMI) | 4 to 8 weeks prior surgery
  Also called the glucose management indicator (GMI) will be calculated from glucose measurements assessed with the Freestyle Libre using accepted algorithms.
Mean levels of sensor-measured interstitial glucose concentration | 4 to 8 weeks prior surgery
  The average glucose values over the past 2 weeks calculated by the freestyle libre,in mmol/l
Glycaemic variability (GV) | 4 to 8 weeks prior surgery
  Glycaemic variability (GV) refers to swings in blood glucose levels. It alludes to blood glucose oscillations that occur throughout the day, including hypoglycemic periods and postprandial increases, as well as blood glucose fluctuations that occur at the same time on different days. The glycaemic variability will be expressed as standard deviation, coefficient of variation, high blood glucose index and low blood glucose index.
Clinical outcomes | 4 to 8 weeks prior surgery
  Clinical outcomes (infections, use of medication including antibiotics, analgetics, insulin (units) and other blood glucose lowering drugs, ICU days, duration of admission) during hospitalization after the VITAAAL intervention via electronic health record data, checked with the patient.
Medication usage | 4 to 8 weeks prior surgery
  Glucose-lowering medication usage at the start and end of the intervention via electronic health record data, checked with the patient.
Blood pressure | 4 to 8 weeks prior surgery
  Blood pressure will be measured during baseline visit
Peripheral neuropathy | 4 to 8 weeks prior surgery
  Peripheral neuropathy will be evaluated with the touch test as part of regular care. This test is performed by pricking the monofilament under the big, middle and small toes of both feet. If the patient does not feel 2 or more of these pricks, this is diagnosed as having peripheral neuropathy.
HbA1c | 4 to 8 weeks prior surgery
  HbA1c values are obtained from blood samples that are taken as part of regular care from the patient record.
Physical activity | 4 to 8 weeks prior surgery
  Physical activity will be assessed using the Fitbit or using the manually entered log-data in the Diameter. Steps per minute assessed with de Fitbit will be used provide information on levels of physical activity. In addition, these data can be used to calculate other activity parameters (e.g., moderate to vigorous physical activity bouts, sedentary behavior, step cadence and peak activity index). To this purpose, scripts in Matlab have previously been developed and tested extensively. Steps per minute and total minutes of moderate to vigorous per week will be used to analyse the intervention effects.
Nutritional behavior | 4 to 8 weeks prior surgery
  Nutritional behavior will be assessed using the food diary in the Diameter. The Diameter logs (number of days logged, and mean number of logs per day), the eaten products at that time and nutritional components (carbohydrates, fat, protein, sugar and kilocalories). To assess the intervention effects, the mean number of carbohydrates, fat, protein, sugar and kilocalories per day will be used. Patients are asked to fill in the food diary for 4 days each week including 2 days in the weekend, as 4 days are required to be able to measure variety in carbohydrabe intake.
Treatment adherence | 4 to 8 weeks prior surgery
  Treatment adherence will be assessed using de Beliefs about Medicines Questionnaire (BMQ). The BMQ consists of 19 items and comprises 2 sections: the BMQ-Specific which assesses representations of medication prescribed for personal use. The score for each subscale is between 5 and 20.
Self-efficacy | 4 to 8 weeks prior surgery
  Self-efficacy will be assessed with all 20 items of the Diabetes Management Self-Efficacy scale for patients with T2DM (DMSES) using a 5-point Likert scale (1 probably not - 5 definitely yes).
Self-management | 4 to 8 weeks prior surgery
  Self-management using the Patient Activation Measure (PAM) a 100-point quantifiable scale determining patient engagement in healthcare. It is a 13-item instrument which assesses patient (or consumer) self-reported knowledge, skills and confidence for self-management of one's health or chronic condition. Based on the PAM score patients can be classified into 4 categories ranging from more passive patients who perceived to have minimal control (1) to having perceived to being absolutely capable of managing their disease (PAM 4).
Stages of change | 4 to 8 weeks prior surgery
  Stages of change using the single intem questionnaire Self-Assessment Scales (SAS) Stages of Change. It assess a person's adherence to lifestyle guidelines using 5-point likert scale.
Health-related quality of life | 4 to 8 weeks prior surgery
  Health-related quality of life using the EQ-5D-5L. The EQ-5D-5L is a generic instrument for describing and valuing health. It defines health in terms of 5 dimensions: mobility, self-care, usual activities, pain/comfort, and anxiety/depression. Each dimension has 5 response categories ranging from no problems (1) to extreme problems (5).
fasting glucose | 4 to 8 weeks prior surgery
  HbA1c values are obtained from blood samples that are taken as part of regular care from the patient record.
  total cholesterol, HDL-cholesterol, LDL-cholesterol, triglycerides, liver enzymes and eGFR. Blood data not older than one month before baseline will be used and stored as part of this study if available.
  Morning void urine will be used to monitor the presence of potential diabetes related complications such as kidney failure. Patients will collect morning void urine as part of regular care, which will be sent to the laboratory for analysis and storage. Morning void data will be derived from the patient record and used for analysis. Urine not older than one months before baseline will be used and stored as part of this study if available.
Cholesterol | 4 to 8 weeks prior surgery
  Cholesterol values are obtained from blood samples that are taken as part of regular care from the patient record.
eGFR | 4 to 8 weeks prior surgery
  eGFR values are obtained from blood samples that are taken as part of regular care from the patient record.
Morning void urine | 4 to 8 weeks prior surgery
  Morning void urine will be used to monitor the presence of potential diabetes related complications such as kidney failure. Patients will collect morning void urine as part of regular care, which will be sent to the laboratory for analysis and storage. Morning void data will be derived from the patient record and used for analysis. Urine not older than one months before baseline will be used and stored as part of this study if available.

CONTACTS AND LOCATIONS:
Locations (1):
- Ziekenhuisgroep Twente, Almelo, Overijssel, Netherlands

IPD SHARING:
Plan to Share IPD: No